CLINICAL TRIAL: NCT06121466
Title: Effect of Abdominal Wall Injections on Abdominal Pain
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Sophia Lichenstein-Hill, Assistant Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00024914
Record Dates: First submitted 2023-09-06; First posted 2023-11-08 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Anterior Cutaneous Nerve Entrapment Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Abdominal wall injections for abdominal wall pain (Experimental): Patients with abdominal pain who are suspected of having abdominal wall pain.
  Interventions: Drug: Abdominal wall injections with lidocaine 2%

INTERVENTIONS:
Drug: Abdominal wall injections with lidocaine 2% — Injections will be administered for patient who are identified as having abdominal wall pain.

SUMMARY:
This is a prospective cohort study of outpatient adults with chronic abdominal wall pain receiving abdominal wall injections, as part of their usual care, with lidocaine. Subjects will be recruited at the outpatient gastroenterology clinic at OHSU.

DETAILED DESCRIPTION:
This is a prospective cohort study of outpatient adults with chronic abdominal wall pain who receive abdominal wall injections with lidocaine at an academic medical center. Thirty patients will be enrolled. A baseline assessment will include a medical history review and survey administration (Pain Catastrophizing Scale, Psychological Inflexibility in Pain Scale, Patient-Reported Outcomes Measurement Information System-29, Recurrent Abdominal Pain Intensity and Disability scale). Subjects will undergo Quantitative Sensory Testing to measure their pain tolerance and thresholds. The primary outcome to be measured is the change in abdominal wall pain at 1 week, 4 weeks and 12 weeks following the abdominal wall injection, with improvement defined as a 50% reduction in baseline pain score measured using an 11-point numeric scale. Data analysis will consist of basic summary statistics to describe the mean, median, and standard deviation for demographic variables and clinical measures. A one-sample t-test or Wilcoxon test will be used to compare differences in continuous values between time points. Chi-square tests will be used to compare differences in categorical variables. An alpha of 0.05 will be used for all statistical tests. Univariate and multivariate logistic regression will be used to assess for factors associated with pain reduction.

ELIGIBILITY:
Inclusion Criteria:

* Localized abdominal wall pain
* Average daily pain (7-day recall) ≥ 3 on a scale of 0-10
* Suspected abdominal wall etiology for abdominal pain
* Positive Carnett's sign or pain near an incisional site
* 18 years of age or older

Exclusion Criteria:

* Suspected visceral etiology for the abdominal pain
* Severe allergy to lidocaine
* Unwillingness or inability to provide informed consent
* Low probability of follow-up
* Abdominal wall hernia noted at the point of pain
* History of trigger point injections for abdominal pain
* Bleeding disorder
* Pregnancy, incarceration or decisionally impaired

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
1) To measure the change in abdominal wall pain 1-week, 1-month and 3-months following abdominal wall injections, with improvement defined as a 50% reduction in baseline pain score measured using an 11-point numeric scale. | 12 weeks
  Improvement is defined as a 50% reduction in baseline pain score measured using an 11-point numeric scale where 0 is no pain and 10 is the worst pain the patient has every felt.
2) To determine patient characteristics, such as pain catastrophizing, associated with a response to abdominal wall injection | 12 weeks
  This will be measured by the following:
  Pain Catastrophizing Scale (PCS):
  Each question is rated on a scale of 0 to 4, where 0 is no catastrophizing, and 4 is significant catastrophizing.
2) To determine patient characteristics, such as patient reported functional status, pain status, and global estimate status; associated with a response to abdominal wall injection | 12 weeks
  This will be measured by the following:
  Routine Assessment of Patient Index Data (RAPID) Questionnaire:
  Assessing patient-reported measures of function, pain, and patient global estimate status. First set of items are rated on a 4-point scale, ranging from 0 to 3, where higher scores indicate lower functioning. Second set of items are rated on a scale from 0 to 10 where the higher the number the more pain the person is experiencing. The third set is rated on a scale from 0 to 10 where 10 is the poorest overall status.
2) To determine patient characteristics, within seven health domains, associated with a response to abdominal wall injection | 12 weeks
  This will be measured by the following:
  Patient-Reported Outcomes Measurement Information System-29 Scale:
  Assessing pain intensity using a single 0-10 numeric rating (0 is no pain, 10 is the worst pain ever felt) item and seven health domains.
2) To determine patient characteristics, such as psychological inflexibility, associated with a response to abdominal wall injection | 12 weeks
  Psychological Inflexibility in Pain Scale:
  Items are rated on a 7-point scale, ranging from 1 to 7, where higher scores indicate greater levels of psychological inflexibility.
3) To determine the rate of adverse events associated with abdominal wall injection. | 12 weeks
  Adverse events associated with abdominal wall injections include pain or discoloration at the injection site, a syncopal episode after the injection, allergic reaction to lidocaine or alcohol swab/chloroprep. There is a rare risk for seizures and injury to a muscle.
4) To measure pain thresholds with use of heat, using quantitative sensory testing (QST) in patients receiving abdominal wall injections. | 12 weeks
  This will be measured by the following:
  Heat Pain Threshold and Pain Tolerance :. This task involves applying a series of heat sensations using a heat thermode (TSA-II Air, Medoc) to the subject's dominant inner forearm.
4) To measure pain thresholds with use of temporal summation, using quantitative sensory testing (QST) in patients receiving abdominal wall injections. | 12 weeks
  This will be measured by the following:
  Temporal summation. For assessment of temporal summation (TS), punctate mechanical stimuli will be delivered to the dorsal surface of the dominant hand using a 300-gm nylon monofilament developed by the German Research Network on Neuropathic Pain.
4) To measure pain thresholds with use of pressure thresholds, using quantitative sensory testing (QST) in patients receiving abdominal wall injections. | 12 weeks
  This will be measured by the following:
  Pressure pain threshold. Pressure pain threshold (PPTh) will be assessed via an algometer using pressure pain stimuli delivered to dorsal forearm (distal stimuli) and the trapezius (order counterbalanced).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - OHSU, Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No